CLINICAL TRIAL: NCT02104687
Title: The Influence of Intraoperative Goal-directed Hemodynamic Therapy Based on Cardiac Index Trending on the Volume of Intraoperatively Administered Fluids and Vasoactive Agents in Comparison to Standard Pressure Monitoring in Patients Undergoing Major Elective Abdominal Surgery
Brief Title: Intraoperative Haemodynamic Optimization Comparing Flow and Pressure Parameters
Acronym: Flow-press
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FNO-KARIM-1; SGS05/LF/2014 (Other Grant/Funding Number: Medical Faculty, Ostrava University)
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Major Abdominal Surgery; Duodenohemipancreatectomy; Rectal Resection; Extensive Bowel Surgery
Keywords: GTD, goal-directed haemodynamic therapy; CI, cardiac index; MAP, mean arterial pressure; CVP, central venous pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flow (Active Comparator): The Flow therapeutic algorithm will be responsible for adjustment of intraoperative interventions - volumotherapy and administration of vasoactive drugs, with the aim to maintain the CI value >2.5 l/m/m2 (FTc - flow time <330 ms was chosen as variable defining preload; PV, peak velocity <70 ms-1 will be used as a variable defining contractility; SVR, total systemic vascular resistance between 1000-1800 cdyn.s/cm5m2 will be used as variable defining after load). After the desired values of CI have been obtained, no further increase of therapeutic intervention (fluids, vasoactive drugs) will be performed.
  Interventions: Procedure: Press group
- Press (Active Comparator): The Press therapeutic algorithm will be responsible for adjustment of intraoperative interventions based upon standard pressure parameters and will include volumotherapy and administration of vasoactive drugs, with the aim to maintain the desired values of MAP of 65-105 mmHg and CVP 8-12 mmHg. After the desired values of MAP and CVP have been obtained, no further increase of therapeutic intervention (fluids, vasoactive drugs) will be performed.
  Interventions: Procedure: Flow group

INTERVENTIONS:
Procedure: Flow group — After induction, each patient will obtain Transesophageal Dopplerometry probe (CardioQ) in order to monitor the parameters of CI, FTc, PV and SVR.
  Arms: Press
Procedure: Press group — After induction, the parameters of MAP and CVP will be monitored in each of the patients.
  Arms: Flow

SUMMARY:
The purpose of the study is to confirm the hypothesis that flow treatment algorithm based on cardiac index trending by transesophageal Dopplerometry would result in reduced complications and reduced length of hospital stay in major abdominal surgery patients, when compared to patients treated with press treatment algorithm.

DETAILED DESCRIPTION:
Despite standardisation of intraoperative care provided for risk surgery patients, the preoperative mortality remains higher than expected. The aim of the goal-directed heamodynamic therapy (GDT) is to improve the altered cardiovascular function and to reach the desired intraoperative values of oxygen supply (DO2) and cardiac index (CI). Standard haemodynamic measurements, such as heart rate (HR), mean arterial pressure (MAP) and central venous pressure (CVP) remain relatively unchanged despite reduced blood flow. However, GTD is able to detect early hypo perfusion abnormalities. The aim of goal-directed heamodynamic therapy, based on the titration of fluids and vasoactive drugs to physiological flow-related end points is to reduce perioperative complications, perioperative morbidity and mortality. We hypothesise, that following this treatment regimen results in reduced postoperative complications (primary endpoint) and reduced length of hospital stay (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and above
* anticipated duration of surgery more than 120 minutes
* estimated blood loss exceeding more than 15% of blood volume
* American Society of Anesthesiology (ASA) classification 2 or 3
* indication for an arterial line and central venous catheter

Exclusion Criteria:

* pregnant or lactating women
* age below 21 years of age
* emergency surgery
* American Society of Anesthesiology (ASA) classification 1
* sepsis and septic shock
* severe cardiac arrhythmias
* patients with pathology or intervention on oesophagus

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pre-defined postoperative complications for up to 28 days after surgery | 24 months
  The followed postoperative complications include infectious, respiratory, cardiovascular, abdominal, renal complications, massive postoperative bleeding and preoperative death.

SECONDARY OUTCOMES:
The length of hospitalization | 24 months
  Length of hospital stay will be obtained from the patient record.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Szturz, MD, Ph.D., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia

REFERENCES:
- [Background] Shoemaker WC, Appel PL, Kram HB. Hemodynamic and oxygen transport responses in survivors and nonsurvivors of high-risk surgery. Crit Care Med. 1993 Jul;21(7):977-90. doi: 10.1097/00003246-199307000-00010. PMID 8319478
- [Background] Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesth Analg. 2011 Jun;112(6):1392-402. doi: 10.1213/ANE.0b013e3181eeaae5. Epub 2010 Oct 21. PMID 20966436